CLINICAL TRIAL: NCT05557240
Title: Clinical Study on the Effect of Neoantigens on the Therapeutic Efficacy and Intestinal Microbiota in Patients With Newly Diagnosed Glioma
Brief Title: Neoantigens Phase I Trial in Newly Diagnosed Glioblastoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Hangzhou NeoVax Biotechnology Co. Ltd. (Industry)
Responsible Party: Principal Investigator, LiangGao, Neurosurgery department, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10247
Record Dates: First submitted 2022-09-25; First posted 2022-09-27 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Glioma, Malignant; Antigen-specific Vaccines; Individualized Treatment
MeSH Terms: conditions — Glioma | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeoPep Vaccine1and 2 plus polyICLC concurrent to TMZ (Experimental)
  Interventions: Drug: NeoPep Vaccine1 plus Poly-ICLC; Drug: NeoPep Vaccine2 plus Poly-ICLC

INTERVENTIONS:
Drug: NeoPep Vaccine1 plus Poly-ICLC — NPVAC1： NPVAC1 drug products are composed of 5 peptides from the HCMV warehouse， NPVAC1 vaccine will be applied before maintenance TMZ cycles after completion of chemoradiation therapy (CRT). Beginning on day 14 before the first maintenance TMZ cycle, patients will receive 7 vaccinations with NPVAC1 drug products during 6 weeks. 400 μg per peptide per vial are used.
  Poly-ICLC:
  Poly-ICLC（500ug）will be used as immunomodulator with all vaccinations.
  Other Names: NPVAC1+Poly-ICLC
Drug: NeoPep Vaccine2 plus Poly-ICLC — NPVAC2： NPVAC2 will be ready for use 2 months after enrollment, as these peptides have to be newly synthesized for each patient following identification of the mutanome and corresponding mutated peptides in the HLA ligandome. NPVAC2 drug products are composed 20 peptides de novo synthesized for an individual patient. Patients will be repeatedly vaccinated with NPVAC2 drug products beginning on day 33 of the 6 maintenance TMZ cycle.Patients will receive 9 vaccinations within 12 weeks. 400 μg per peptide per vial are used.
  Poly-ICLC:
  Poly-ICLC（500ug）will be used as immunomodulator with all vaccinations.
  Other Names: NPVAC2+Poly-ICLC

SUMMARY:
The primary objective of this study is to assess the safety and tolerability, feasibility of the NeoPep Vaccine in newly diagnosed glioblastoma (GB) patients.

DETAILED DESCRIPTION:
This is a signelcenter, open-label, single arm, first-in-human phase I trial to investigate the safety, feasibility and immune response of the novel NeoPep Vaccine in patients with newly diagnosed GB.

Primary Endpoints:

Determine the safety and tolerability profile of NeoPep Vaccine1and 2 when administered with immunomodulators and Stupp standard treatment

Secondry Endpoints:

1. Descriptive analysis of induced T-cell immune responses after vaccinations with NeoPep Vaccine1and 2 drug products plus immunomodulators and Stupp standard treatment.
2. Overall survival with NeoPep Vaccine1 and 2 plus immunomodulator in newly diagnosed glioma in patients treated with standard Stupp.
3. Progression-free survival with NeoPep Vaccine1 and 2 plus immunomodulator in newly diagnosed glioma in patients treated with standard Stupp.

After the standard chemoradiotherapy with TMZ has been completed, Vaccination was initiated 14 days before the first maintenanceTMZ cycle. It starts with the first NeoPep Vaccine1, followed by additional NeoPep Vaccine2 at a later time point and ends with the Last Endpoint Evaluation Visit (LEEV) of a patient.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of subject to understand and the willingness to sign written informed consent for study participation;
2. Patients with newly diagnosed high-grade glioma confirmed by histopathological and imaging evaluation;
3. Gross total resection (as defined by less than 1 cm2 residual tumor mass on the largest perpendicular axes in post-operative scan taken within 48 h post-surgery; standard MRI conformable to the present national and international guidelines is sufficient)；
4. At least 0.5 g tumor tissue freshly cryopreserved during surgery，and could provide adequate amounts of PBMC；
5. Patient is a candidate for and willing to receive standard CRT with TMZ followed by maintenance TMZ cycles;
6. Age 18-70;
7. Life expectancy > 9 months;
8. KPS≥70;
9. Sufficient tumor tissue samples and peripheral blood samples can be obtained for sequencing analysis, or whole exome sequencing and RNA sequencing of tumor tissue samples and peripheral blood samples have been obtained, and the sequencing data meet the prediction requirements;
10. Consent of women and men of reproductive age to use adequate and effective contraception during clinical trials;
11. Normal laboratory values for hematology, liver and renal function (serum creatinine).In detail the following values apply as inclusion criteria:

    1. White blood cell count (WBC) ≥3.0×109/L；
    2. Absolutely neutrophil count≥1.0×109/L；
    3. Platelet count≥80×109/L；
    4. Hemoglobin content≥90g/L；
    5. Serum creatinine≤1.5 ULN or Creatinine clearance rate≥40 mL/min;
    6. TBil(total bilirubin)≤1.5 x ULN;
    7. Aspartic transaminase(AST)≤2.5x ULN or Alanine aminotransferase（ALT）≤2.5x ULN；Patients with liver metastases must have ≤5x ULN;
    8. Blood coagulation function :INR≤1.5x ULN；pT and APTT≤1.5x ULN;
    9. Urine protein< 2 +;if Urine protein≥2+,24-hour urinary protein must be less than 1g.

Exclusion Criteria:

1. Patients treated with immunosuppressive agents (e.g., cyclosporin CsA, tacrolimus, rapamycin, azathioprine, etc.) within the previous month; Other immunotherapy within 3 months;
2. History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within the last 5 years unless the patient has been disease-free for 5 years;
3. Participated in other clinical trials within 30 days prior to screening;
4. Have a history of severe allergy or allergic constitution;
5. Patients who have undergone splenectomy;
6. Persons with primary or secondary immunodeficiency diseases (e.g. AIDS);Patients with autoimmune diseases;
7. Patients who received multiple oral, intramuscular, or intravenous corticosteroids within 30 days before the first dose; However, patients who received a single oral, intramuscular, or intravenous dose of dexamethasone of 5mg or less (or another hormone of equivalent potency) 14 days before the first dose were allowed; Allow inhaled corticosteroids to treat respiratory insufficiency (e.g., chronic obstructive pulmonary disease), or topical steroids;
8. Patients with uncontrollable seizures, central nervous system disorders, or psychotic loss of cognition;
9. Uncontrolled central nervous system metastases;
10. Patients had a history of chronic alcohol or drug abuse in the 6 months before screening;
11. With unstable systemic disease, such as active infection, liver cirrhosis, chronic renal failure, severe chronic pulmonary disease, unstable hypertension, unstable angina pectoris, congestive heart failure, myocardial infarction within one year, etc. ;
12. According to this procedure, the number of candidate neoantigens that can be used to make personalized vaccines is less than 20;
13. The investigator did not consider it appropriate to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-02-12 (Estimated); Study Completion 2025-08-12 (Estimated)

PRIMARY OUTCOMES:
Safety and toleration | Continously for about 40 weeks plus follow-up
  Determine the safety and tolerability profile of NeoPep Vaccine1and 2 when administered with immunomodulators and Stupp standard treatment

SECONDARY OUTCOMES:
T-cell immune response | till 24 months of vaccination
  Descriptive analysis of induced T-cell immune responses after vaccinations with NeoPep Vaccine1and 2 drug products plus immunomodulators and Stupp standard treatment.
Overall survival(OS) | till 24 months of vaccination
  Overall survival with NeoPep Vaccine1 and 2 plus immunomodulator in newly diagnosed glioma in patients treated with standard Stupp.
Progression-free survival（PFS） | till 12 months of vaccination
  Progression-free survival with NeoPep Vaccine1 and 2 plus immunomodulator in newly diagnosed glioma in patients treated with standard Stupp.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Gao, Phd, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No